CLINICAL TRIAL: NCT00672243
Title: Phase II Trial of Erlotinib Plus Sirolimus for Patients With Recurrent Malignant Glioma Multiforme
Brief Title: Ph II Erlotinib + Sirolimus for Pts w Recurrent Malignant Glioma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Genentech, Inc. (Industry); OSI Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00000345
Record Dates: First submitted 2008-01-29; First posted 2008-05-06 (Estimated); Results first posted 2013-04-04 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-07

CONDITIONS: Glioblastoma; Gliosarcoma
Keywords: GBM; Brain tumor; Erlotinib; Sirolimus; Glioblastoma multiforme; Glioblastoma; Gliosarcoma3; Tarceva; Rapamune
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Brain Neoplasms | interventions — Erlotinib Hydrochloride; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Erlotinib + Sirolimus (Experimental): Erlotinib & sirolimus on a daily dosing schedule on a 28-day cycle. Dosing was 150 mg of erlotinib and 5mg of sirolimus for patients not on concurrent Cytochrome P450, family 3 (CY3PA)-inducing anti-epileptics (EIAEDS) and 400 mg of erlotinib and 10 mg of sirolimus for patients on concurrent EIAEDS.
  Interventions: Drug: Erlotinib + sirolimus

INTERVENTIONS:
Drug: Erlotinib + sirolimus — Erlotinib & sirolimus on a daily dosing schedule on a 28-day cycle. Dosing was 150 mg of oral erlotinib and 5mg of oral sirolimus for patients not on concurrent CY3PA-inducing anti-epileptics (EIAEDS) and 400 mg of oral erlotinib and 10 mg of oral sirolimus for patients on concurrent EIAEDS.
  Other Names: sirolimus - Rapamune; erlotinib - Tarceva - OSI-774

SUMMARY:
Primary objective:

To determine the 6-month progression free survival of patients with recurrent glioblastoma multiforme (GBM) treated with Erlotinib plus Sirolimus.

Secondary objectives:

To further define the safety and tolerability of Erlotinib plus Sirolimus when administered to patients with recurrent GBM; and to evaluate progression free survival, radiographic response and overall survival of patients with recurrent GBM treated with Erlotinib plus Sirolimus.

DETAILED DESCRIPTION:
The primary objective of this study will be to determine the 6-month progression free survival of patients with recurrent GBM treated with Erlotinib plus Sirolimus.

This is an exploratory, single-arm, phase II study designed to assess the anti-tumor activity of a combinatorial regimen consisting of Erlotinib plus Sirolimus among patients with recurrent GBM. The combinatorial regimen of Erlotinib plus Sirolimus is rationally designed to simultaneously inhibit upstream (EGFR) and downstream (mTOR) mediators of Phosphatidylinositide 3-kinase/Protein Kinase B (PI3/AKT) signaling. In a recently completed phase I study, we determined that an EGFR inhibitor (Gefitinib) can be safely combined with Sirolimus at dose levels that are routinely used in the monotherapy setting. Therefore, the primary endpoint of this study is the probability of progression-free survival at 6 months among recurrent GBM patients treated with standard doses of Erlotinib plus Sirolimus. An important secondary objective is to further assess the safety of Erlotinib and Sirolimus for patients with recurrent GBM.

ELIGIBILITY:
Inclusion Criteria:

* Pts have confirmed diagnosis of recurrent primary WHO grade IV malignant glioma (MG). Pts w recurrent disease whose diagnostic pathology confirmed GBM will not need re-biopsy. Pts w prior low-gr glioma / anaplastic glioma are eligible if histologic assessment demonstrates transformation to GBM
* Age >18 yrs
* Interval of >2 wk between prior surgical resection
* Interval of >12 wks between prior external-beam radiation therapy (XRT) unless there is either: histopathologic confirmation of recurrent tumor; new enhancement on MRI outside of XRT treatment field; / progressive radiographic changes after XRT/temo as well as after adjuvant, post-XRT temo
* Interval of >4 wks between chemo & enrollment on protocol unless: unequivocal evidence of tumor progression; & pt has recovered fully from all toxicity associated w prior surgery, XRT/chemo. Pts treated w chemo agents such as VP-16 who would normally be retreated after shorter intervals may be treated at usual starting time even if <4 wks from last prior dose chemo
* Karnofsky performance score >= 70 percent
* Hematocrit >29 percent, absolute neutrophil count (ANC) >1,500 cells/microliter, platelets >100,000 cells/microliter
* Serum creatinine <1.5 mg/dl, serum glutamic oxaloacetic transaminase (SGOT) & bilirubin <1.5 x upper limit of normal (ULN); fasting plasma triglyceride & cholesterol < gr1
* For pts on corticosteroids, dose should not be increasing for >7 days prior to baseline Gd-MRI of brain if medically appropriate
* Pts in enzyme inducing antiepileptic drug cohort must be on stable dose of p450-inducing EIAED for >2 wks. Pts in non-EIAED cohort must not receive any p450-EIAED for >2 wks prior to & during participation in trial
* Signed informed consent approved by Institutional Review Board (IRB) prior to pt entry
* If sexually active, pts will take contraceptive measures for duration of treatments & for 3 months following discontinuation of Erlotinib
* Pts who have had prior bevacizumab are eligible however interval of >6 weeks must have elapsed since their last dose

Exclusion Criteria:

* Prior mammalian target of rapamycin (mTOR) directed therapy
* Prior epidermal growth factor receptor (EGFR)-directed therapy
* Female pts are pregnant/breast feeding, or adults of reproductive potential not employing effective method of birth control. Women of childbearing potential must have negative serum pregnancy test <72 hours prior to administration of Erlotinib
* Co-medication that may interfere w study results
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring IV antibiotics, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, hyperlipidemia not controlled w medication, psychiatric illness/social situations that would limit compliance w study requirements,/disorders associated w significant immunocompromise
* Acute/chronic liver disease
* Impairment of GI function/GI disease that may significantly alter absorption of Erlotinib
* Pts who have received investigational drugs <4 wks prior to entry on study or who have not recovered from toxic effects of such therapy
* Pts who have received biologic, immunotherapeutic/cytostatic agents <1 wk prior to entry on study/have not recovered from toxic effects of such therapy
* Pt is <5 yrs free of another primary malignancy except: if other primary malignancy is not currently clinically significant/requiring active intervention,/if other primary malignancy is basal cell skin cancer/cervical carcinoma in situ. Existence of any other malignant disease is not allowed
* Pts have had any surgery other than resection of brain tumor <2 wks prior to entry on study/have not recovered from side effects of such therapy
* Pts unwilling to/unable to comply w protocol
* Pts w acute/chronic renal insufficiency/those w acute renal insufficiency of any severity due to hepato-renal syndrome/in peri-operative liver transplantation period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-04; Primary Completion 2008-09 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Reardon, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

REFERENCES:
- [Result] Reardon DA, Desjardins A, Vredenburgh JJ, Gururangan S, Friedman AH, Herndon JE 2nd, Marcello J, Norfleet JA, McLendon RE, Sampson JH, Friedman HS. Phase 2 trial of erlotinib plus sirolimus in adults with recurrent glioblastoma. J Neurooncol. 2010 Jan;96(2):219-30. doi: 10.1007/s11060-009-9950-0. Epub 2009 Jun 28. PMID 19562254
- See also: The Preston Robert Tisch Brain Tumor Center at DUKE — http://www.cancer.duke.edu/btc/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled between May 2007 and March 2008 at the Preston Robert Tisch Brain Tumor Center at Duke.
Pre-assignment Details: Patients were excluded for any of the following: prior therapy with either an EGFR or mTOR antagonist; uncontrolled intercurrent illness including active infection, symptomatic congestive heart failure, unstable angina, grade 3 or greater hyperlipidemia or significant gastrointestinal, renal or liver disease, pregnancy or nursing
Groups:
- Erlotinib + Sirolimus: Erlotinib & sirolimus on a daily dosing schedule on a 28-day cycle. Dosing was 150 mg of erlotinib and 5mg of sirolimus for patients not on concurrent Cytochrome P450, family 3, subfamily A (CY3PA)-inducing anti-epileptics (EIAEDS) and 400 mg of erlotinib and 10 mg of sirolimus for patients on concurrent EIAEDS.
Period: Overall Study
Arm/Group | Erlotinib + Sirolimus
Started | 32
Completed | 32
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Erlotinib + Sirolimus: Erlotinib & sirolimus on a daily dosing schedule on a 28-day cycle. Dosing was 150 mg of erlotinib and 5mg of sirolimus for patients not on concurrent CY3PA-inducing anti-epileptics (EIAEDS) and 400 mg of erlotinib and 10 mg of sirolimus for patients on concurrent EIAEDS.
Arm/Group | Erlotinib + Sirolimus
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 7
Age, Customized [Median (Full Range); unit: years] | 54 [40 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 25
Karnofsky Performance Scale (KPS) [Number; unit: participants] — Karnofsky Performance Scores (KPS) range from 0-100 (100=Normal, no complaints; no evidence of disease; 90=Able to carry on normal activity; minor signs or symptoms of disease; 80=Normal activity with efforts; some signs or symptoms of disease; 70=Cares for self; unable to carry on normal activity or to do active work. Scores between intervals are possible.
  participants
    100 | 4
    90 | 13
    85 | 1
    80 | 9
    70 | 5
Received prior bevacizumab [Number; unit: participants]
  Yes | 9
  No | 23
Enzyme-inducing anti-epileptic drug (EIAED) status [Number; unit: participants]
  Not receiving EIAEDs | 24
  Receiving EIAEDs | 8

OUTCOME MEASURES:

1. Primary Outcome: 6-month Progression-free Survival (PFS)
Description: Percentage of participants surviving six months from the start of study treatment without progression of disease. PFS was defined as the time from the date of study treatment initiation to the date of the first documented progression according to the Macdonald criteria, or death due to any cause. Progression based on Macdonald criteria is defined as a ≥ 25% increase in the sum of the products of perpendicular diameters of enhancing lesions; any new lesion; or clinical deterioration.
Time Frame: 6 months
Population: Intent to treat (ITT)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Erlotinib + Sirolimus
Number analyzed (Participants) | 32
percentage of participants | 3.1 [0.2 to 13.7]

2. Secondary Outcome: Median Progression Free Survival (PFS)
Description: Time in weeks from the start of study treatment to the date of first progression according to Macdonald criteria, or to death due to any cause. Patients alive who had not progressed as of the last follow-up had PFS censored at the last follow-up date. Median PFS was estimated using a Kaplan-Meier curve. Progression based on Macdonald criteria is defined as a ≥ 25% increase in the sum of the products of perpendicular diameters of enhancing lesions; any new lesion; or clinical deterioration.
Time Frame: 2 years
Population: Intent to treat (ITT)
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Erlotinib + Sirolimus
Number analyzed (Participants) | 32
weeks | 6.9 [3.9 to 11]

3. Secondary Outcome: Median Overall Survival (OS)
Description: Time in weeks from the start of study treatment to date of death due to any cause. Patients alive at last follow-up are censored as of that follow-up date. Median OS was estimated using a Kaplan-Meier curve.
Time Frame: 2 years
Population: Intent to treat (ITT)
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Erlotinib + Sirolimus
Number analyzed (Participants) | 32
weeks | 33.8 [21.9 to 53.6]

4. Secondary Outcome: Best Radiographic Response
Description: Best radiographic response per modified Macdonald criteria. Complete response: disappearance of all enhancing tumor, no new lesions, and no steroids or only maintenance doses. Partial response: ≥ 50% reduction in the products of the perpendicular diameters of all enhancing lesions, no new lesions, & steroids must be at a stable/decreasing dose. Stable disease: does not qualify for complete or partial response or progression & is stable clinically. Progression: ≥ 25% increase in the sum of the products of perpendicular diameters of enhancing lesions, any new lesion or clinical deterioration.
Time Frame: 2 years
Population: Intent to treat (ITT)
Measure: Number; unit: participants
Arm/Group | Erlotinib + Sirolimus
Number analyzed (Participants) | 32
participants
  Complete Response | 0
  Partial Response | 0
  Stable Disease | 15
  Progressive Disease | 16
  Not evaluable | 1

5. Secondary Outcome: Number of Participants Experiencing a ≥ Grade 3, Treatment-related, Non-hematologic Toxicity.
Description: Number of participants experiencing a ≥ grade 3, treatment-related, non-hematologic toxicity.
Time Frame: 2 years
Population: Intent to treat (ITT)
Measure: Number; unit: participants
Arm/Group | Tarceva and Rapamycin
Number analyzed (Participants) | 32
participants | 15

ADVERSE EVENTS:
Time Frame: 2 years
Description: All adverse events were entered using Common Toxicology Criteria (CTC) v. 3.0, but were converted to CTC v. 4.0 for entry into ClinicalTrials.gov
Arm/Group | Tarceva and Rapamycin
Serious Adverse Events (participants affected / at risk) | 4/32
Other Adverse Events (participants affected / at risk) | 26/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tarceva and Rapamycin (N=32)
Abdominal pain (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Fever (General disorders) | 2
Skin infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Platelet count decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tarceva and Rapamycin (N=32)
Anemia (Blood and lymphatic system disorders) | 3
Blurred Vision (Eye disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Diarhhea (Gastrointestinal disorders) | 14
Mucositis oral (Gastrointestinal disorders) | 12
Nausea (Gastrointestinal disorders) | 3
Rectal pain (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 11
Fever (General disorders) | 4
Alanine aminotransferase increase (Investigations) | 12
Aspartate aminotransferase increased (Investigations) | 11
Blood bilirubin increased (Investigations) | 3
Cholesterol high (Investigations) | 18
Investigations-Other, specify: Low Total Protein (Investigations) | 2
Neutrophil count decreased (Investigations) | 3
Platelet count decreased (Investigations) | 12
Weight loss (Investigations) | 3
White blood cell decreased (Investigations) | 7
Anorexia (Metabolism and nutrition disorders) | 5
Hyperglycemia (Metabolism and nutrition disorders) | 11
Hypermagnesemia (Metabolism and nutrition disorders) | 2
Hypernatremia (Metabolism and nutrition disorders) | 2
Hypertriglyceridemia (Metabolism and nutrition disorders) | 11
Hypoalbuminemia (Metabolism and nutrition disorders) | 11
Hypocalcemia (Metabolism and nutrition disorders) | 4
Hypokalemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 3
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2
Ataxia (Nervous system disorders) | 10
Cognitive disturbance (Nervous system disorders) | 6
Depressed level of consciousness (Nervous system disorders) | 4
Dysphasia (Nervous system disorders) | 4
Headache (Nervous system disorders) | 4
Memory impairment (Nervous system disorders) | 6
Peripheral motor neuropathy (Nervous system disorders) | 7
Peripheral sensory neuropathy (Nervous system disorders) | 6
Tremor (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 3
Confusion (Psychiatric disorders) | 7
Insomnia (Psychiatric disorders) | 5
Urinary incontinence (Renal and urinary disorders) | 2
Reproductive system and breast disorders-Other, specify: Sexual dysfunction (Reproductive system and breast disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 18
Investigations-Other, specify: BUN High (Investigations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes